CLINICAL TRIAL: NCT00724295
Title: PEG Intron/REBETOL Combination Therapy Special Investigation -Investigation on the Safety and Efficacy of PegIntron and REBETOL Combination Therapy in Patients With Chronic Hepatitis C-
Brief Title: Safety and Efficacy of PegIntron and Rebetol Combination Therapy in Patients With Chronic Hepatitis C in Japan (Study P04505)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04505
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm 1: Overall study population
  Interventions: Drug: peginterferon alfa-2b; Drug: ribavirin

INTERVENTIONS:
Drug: peginterferon alfa-2b — PegIntron powder (reconstituted) administered in accordance with approved labeling; Subcutaneous injection of 1.5 ug/kg once weekly for 48 weeks.
  Other Names: PegIntron; SCH 54031
Drug: ribavirin — Rebetol capsule administered orally twice daily in accordance with approved labeling (weight based dosing). Dosing duration 48 weeks.
  Other Names: Rebetol; SCH 18908

SUMMARY:
This is a post-marketing surveillance of patients with chronic hepatitis C treated with PegIntron and Rebetol combination therapy in clinical practice in Japan. The objective of the study is to evaluate the safety and efficacy of the combination therapy. The study will also compare the safety profile of the combination therapy among elderly patients and younger patients.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

ELIGIBILITY:
Inclusion Criteria:

Patients with chronic hepatitis C.

* Patients are serogroup 1(genotype I (1a) or II (1b)).
* The HCV-RNA level in the blood is more than 10^5 IU/mL by RT-PCR method, or 1Meq./mL by b-DNA method

Exclusion Criteria:

* Patients with a history of hypersensitivity to test drugs or other interferon preparations
* Patients with a history of hypersensitivity to biological products, such as vaccines
* Patients being treated with Shosaikoto
* Patients with autoimmune hepatitis
* Pregnant women, women who may be pregnant, and nursing mothers
* Patients with a history of hypersensitivity to any component of this drug or other nucleoside analogs (aciclovir, ganciclovir, vidarabine, etc.)
* Patients with difficult-to-control cardiac disease (eg, myocardial infarction, cardiac failure, arrhythmia)
* Patients with hemoglobinopathies (eg, thalassemia, sickle-cell anemia)
* Patients with chronic renal failure or renal function disorder with creatinine clearance of <=50 mL/min
* Patients with or a history of severe psychiatric condition such as severe depression, suicidal ideation or suicide attempt
* Patients with serious hepatic dysfunction
* Patients with autoimmune hepatitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic hepatitis C treated with PegIntron and Rebetol combination therapy in the clinical practice at approximately 100 to 200 institutions in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 1077 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Overall incidence of adverse events and adverse drug reactions. | From the time the informed consent is signed and up to 30 days after study completion or discontinuation. Treatment period is 48 weeks with a 24 week post dose followup.
Assessment of trends of adverse drug reactions by patient factors and concomitant medications. Incidence of adverse events (AEs) in the elderly vs younger patients; rates of hematologic AEs; dose reduction and discontinuation rates. | From the time the informed consent is signed and up to 30 days after study completion or discontinuation. Treatment period is 48 weeks with a 24 week post dose followup.
Sustained virologic response rate and improvement of ALT (alanine transaminase). | Assessed at the end-of-treatment and at 24 weeks post-treatment.